CLINICAL TRIAL: NCT06291311
Title: Treatment of Infections of the Cervix Uteri With High- and Low-risk Variants of the Human Papillomavirus Using Non-invasive Physical Plasma
Brief Title: Non-Invasive Plasma Treatment for Cervical Infections: Targeting High- and Low-Risk HPV Variants
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MT_NIPP-HPV_ERBE
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04

CONDITIONS: HPV Infection; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIPP treatment: Treatment with cold physical Plasma
  Interventions: Other: Cold physical Plasma
- Control group: No treatment with cold physical Plasma
  Interventions: Other: Control group

INTERVENTIONS:
Other: Cold physical Plasma — The treatment is administered by either the supervising specialists or assistant doctors at the University Women's Hospital, under their supervision and authorization. It's important to note that the NIPP treatment is designed to be relatively brief, with a duration not exceeding 10-20 minutes.
  Groups: NIPP treatment
Other: Control group — A potential natural healing of the HPV infection will be anticipated
  Groups: Control group

SUMMARY:
This is a prospective, single-center, observational proof-of-principle clinical trial at the Department of Women's Health of the University Hospital Tübingen.

DETAILED DESCRIPTION:
The aim of this study is to investigate the HPV (Human papillomavirus)-eradicating efficacy of NIPP (non-invasive physical plasma) in patients with confirmed HPV infection but without cervical dysplasia. Another objective is to examine cellular/molecular/immunological effects of NIPP on the cervix through molecular biological methods following in-vivo treatment. Tissue samples will be obtained at defined intervals via minibiopsy, and analyses will be conducted using molecular biological, histological, and microscopic methods, potentially in collaboration with other research institutes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for NIPP treatment

  * Age ≥ 18 years
  * mRNA or DNA-based virus detection by smear (also external findings)
  * Clearly visible transformation zone of the cervix and margins of the lesions corresponding to T1/T2
  * Written informed consent to participate in the study
* Inclusion criteria for control group

  * Age ≥ 18 years
  * Swab-based mRNA or DNA-based virus detection (also external findings)
  * Clearly visible transformation zone of the cervix corresponding to T1/T2
  * Written informed consent to participate in the study

Exclusion criteria:

The following exclusion criteria apply to both groups of patients (NIPP treatment and control group).

* Transformation zone not fully visible
* Evidence of invasive disease
* Serious cardiovascular diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients aged 18 and over from the dysplasia clinic of the University Women's Hospital Tübingen who have been diagnosed with an infection of the cervix uteri involving both high- and low-risk HPV viruses.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HPV eradication rate | 3-6 months
  In the following intervention study, participants will be tested for HPV infection before and after NIPP treatment.

SECONDARY OUTCOMES:
Correlation of HPV Genotyping | During the study (12-24 months)
  HPV genotyping is crucial for identifying specific viral strains. Correlation studies will be performed via obtained datasets and the application of statistical methods to identify associations among different HPV genotypes. The findings from this study will contribute to our understanding of the virus, guide health interventions, and improve clinical management strategies related to HPV infections.
HPV-Quality-of-Life (HPV-QoL) | During the study (12-24 months)
  The HPV-Quality-of-Life (HPV-QoL) questionnaire is developed to determine the impact of HPV infection and related interventions on women health-related quality-of-life.
Tissue Tolerance and Compatibility of NIPP Treatment | During the study (12-24 months)
  Cold plasma generates reactive oxygen and nitrogen species, electric fields, and other biologically active components that can interact with biological tissues. Assessing tissue tolerance and compatibility will be crucial for ensuring the safety and effectiveness of cold plasma treatment.
Detection of Intracellular Molecular Plasma Mechanisms | During the study (12-24 months)
  The detection of intracellular molecular plasma mechanisms refers to the identification and study of processes and mechanisms that take place within cells through the interaction with so-called plasma, especially cold plasma. The detection of intracellular molecular plasma mechanisms refers to the identification and study of processes that take place within cells through the interaction with plasma, especially cold plasma. Interaction of cold plasma with cellular mechanisms will be studied via routine molecular biological methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weiss, Dr. med., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany